CLINICAL TRIAL: NCT04393142
Title: Observational Trial Evaluating the Serologic Status of Household Contacts of Patients Diagnosed With COVID-19
Brief Title: Serologic Testing of Household Contacts of Confirmed Cases of COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Head of the Infectious Disease Department, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: IF20-00004
Record Dates: First submitted 2020-04-26; First posted 2020-05-19 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; IgM/IgG antibodies; Intradomestic contacts; IgM/IgG serological tests
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood samples will be obtained by capillary puncture or venipuncture for rapid testing of antibodies against SARS-CoV-2 (IVD COVID-19 IgM/IgG test kit, Singclean).
  Samples will be stored in the laboratory, and discarded at the discretion of the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SARS-CoV-2 has now crossed the 1 million number of cases and tens of thousands of deaths. It´s R0 has been calculated between 2 and 5.7 solely based on clinical symptoms but it is estimated to likely be higher. Serologic evidence of infection has not been analyzed.

DETAILED DESCRIPTION:
Transverse, observational and descriptive study involving household contacts of documented patients with COVID-19 infection: contacts will be invited to participate and a blood sample will be drowned: IgM and IgG qualitative and quantitative measurements will be performed. Demographic data regarding age, comorbidities, calculated time spent before and after the patients diagnosis, isolation practices etc.

ELIGIBILITY:
Inclusion Criteria:

1. Persons over 1 years of age.
2. .Meet COVID-19 confirmed case intradomestic contact definition:

   1. Living in the same home as the patient with SARS-CoV-2 PCR test detected (nasopharyngeal and/or oropharyngeal swab) performed in the Acute Respiratory Infection Diagnostic Unit.
   2. Living in the same home as the patient with a PCR test for SARS-CoV-2 Indeterminate (nasopharyngeal and/or oropharyngeal swab) performed in the Acute Respiratory Infection Diagnostic Unit and that the initial patient has positive IgM/IgG serology for SARS-CoV-2.
3. .Informed Consent.

Exclusion Criteria:

1. .Have fever, cough, pharyngeal pain or clinically have symptoms compatible with COVID-19 at the time of recruitment.
2. .Autoimmune disease, cancer, neutropenia.
3. .Under 1 years of age.
4. .Patients who, in the investigator's opinion, should be excluded from the research protocol.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The intradomiciliary contacts of the patients with a detected SARS-CoV-2 PCR test (nasopharyngeal and / or oropharyngeal swab) performed at the Acute Respiratory Infection Diagnosis Unit between March 2020 and May 2020 will be located: will invite to participate in the study to record their clinical and demographic data and to take serological samples by venipuncture or fingerstick to perform rapid tests for antibodies against SARS-CoV-2 (IVD COVID-19 IgM / IgG test kit, Singclean).
  Informed consent shall be obtained from each person for the collection of samples. The data collected will be captured in an electronic database in Excel.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Identify antibodies | 1 day
  Identify the presence of IgM and IgG antibodies from intradomestic contacts of patients with Polymerase Chain Reaction for detected SARS-CoV-2 .

SECONDARY OUTCOMES:
Determine antibody sensitivity | 1 day
  Determine the sensitivity of IgM and IgG antibody detection by ELISA in direct eastern contacts of patients with PCR for detected SARS-CoV-2.
IgM determination | 1 day
  Determine the presence of IgM antibodies by ELISA in direct eastern contacts of patients with detected SARS-CoV-2 PCR.
IgG determination | 1 day
  Determine the presence of IgG antibodies by ELISA in direct eastern contacts of patients with detected SARS-CoV-2 PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Camacho-Ortiz, MD, Principal Investigator — Hospital Universitario "Dr. Jose Eleuterio Gonzalez, UANL
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Maier HJ, Bickerton E, Britton P. Preface. Coronaviruses. Methods Mol Biol. 2015;1282:v. doi: 10.1007/978-1-4939-2438-7. No abstract available. PMID 25870870
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Patel A, Jernigan DB; 2019-nCoV CDC Response Team. Initial Public Health Response and Interim Clinical Guidance for the 2019 Novel Coronavirus Outbreak - United States, December 31, 2019-February 4, 2020. MMWR Morb Mortal Wkly Rep. 2020 Feb 7;69(5):140-146. doi: 10.15585/mmwr.mm6905e1. PMID 32027631
- See also: "About the Virus." World Health Organization, World Health Organization, 17 Apr. 2020 — http://www.euro.who.int/en/health-topics/health-emergencies/coronavirus-covid-19/novel-coronavirus-2019-ncov
- See also: "Naming the Coronavirus Disease (COVID-19) and the Virus That Causes It." World Health Organization. World Health Organization. Accessed April 17, 2020. — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance/naming-the-coronavirus-disease-(covid-2019)-and-the-virus-that-causes-it
- See also: Johns Hopkins Coronavirus Resource Center." Johns Hopkins Coronavirus Resource Center. Accessed April 17, 2020. — https://coronavirus.jhu.edu/map.html.
- See also: Comparative Accuracy of Oropharyngeal and Nasopharyngeal Swabs for Diagnosis of COVID-19." CEBM. Accessed April 17, 2020. — https://www.cebm.net/covid-19/comparative-accuracy-of-oropharyngeal-and-nasopharyngeal-swabs-for-diagnosis-of-covid-19/.
- See also: 12. Cdc. "Coronavirus Disease 2019 (COVID-19)." Centers for Disease Control and Prevention. Accessed April 17, 2020 — https://www.coronavirus.gov/.